CLINICAL TRIAL: NCT04065685
Title: A Nurse-led Patient-centred Intervention to Increase Written Advance Directives for Outpatients With Progressive Chronic Illnesses: a Randomized Controlled Trial With an Embedded Explanatory Qualitative Study
Brief Title: A Nurse-led Patient-centred Intervention to Increase Written Advance Directives
Acronym: anticip@imad
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19: participants is a population at risk
Sponsor: Katia Iglesias (Other)
Collaborators: School of Health Sciences Geneva (Other); University Hospital, Geneva (Other); Institution genevoise de maintien à domicile (Unknown); High School for Social Work and Health, Lausanne (Unknown); Swiss Academy of Medical Sciences (SAMS) (Other)
Responsible Party: Sponsor-Investigator, Katia Iglesias, Professor HES, University of Applied Sciences of Western Switzerland
Organization: University of Applied Sciences of Western Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: anticip@imad_PC_12/18
Record Dates: First submitted 2019-06-27; First posted 2019-08-22 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Advance Care Planning; Outpatients; Palliative Care

STUDY DESIGN:
Intervention Model Description: a randomised controlled trial with three parallel arms (with a waiting list for the control group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CG (Active Comparator): control group receiving the usual care, the standardized information on anticipated directives
  Interventions: Other: usual care
- IG p+r (Active Comparator): intervention group with patients and her/his relative
  Interventions: Other: serious game named Go Wish
- IG p (Active Comparator): intervention group with patients without relative
  Interventions: Other: serious game named Go Wish

INTERVENTIONS:
Other: serious game named Go Wish — The nurse led intervention Go Wish is composed of 36 cards presenting statements of personal needs, values, and beliefs about end-of-life care. The aim is to decide about what to put into the patient's file as care options and the subsequent appointments to name a potential surrogate or to elaborate ADs.
  Patient and relative (if participating) will meet their nurse twice:
  Session 1: patient the cards in three piles and to rank the ten most important. Session 2 without relative: the nurse reiterates the wishes of care and treatments previously expressed and links them to the state of health and symptoms of the patient and the current treatments and their possible evolution.
  Session 2 with a relative: the relative sort the cards based on his/her beliefs about the patient's expectation.
  Session 3 with a relative: the nurse bring together the patient and his/her relative to discuss the priorities selected independently, identify, and explore the similarities and differences.
  Arms: IG p; IG p+r
Other: usual care — Standardized information on anticipated directives (ADs): the imad nurse are trained to promote AD to clients to help nurses to describe and explain ADs, to identify and to mobilize the required interview condition to promote ADs to clients to facilitate and initiate discussion on ADs
  Arms: CG

SUMMARY:
Background and rationale: Since 2013, with the new Swiss Adult Protection Law, Anticipated Directives (ADs) have been used to identify patients' wills in case they cannot express them later. This instrument is considered to improve care quality, reduce conflicts in decisions between patients, relatives and healthcare teams and utilisation of health resources. Despite their perceived utility, political and institutional campaigns have failed to make ADs common among the population. Discussing life threatening diseases evolution and end-of-life (EOL) issues remains difficult for patients, relatives and professionals. Several interventions were developed to improve advance care planning (ACP) and lead to ADs. However, most of them are cognitively demanding or requiring high levels of literacy. People in 'early stage palliative care' (i.e. with chronic degenerative conditions) could benefit from a simple, adjusted, and acceptable intervention to address the problem outside the hospital setting before the crisis and the appearance of other complications. For a dialogue about EOL to take place, it is necessary to engage in a trustful therapeutic relationship constructed on favourable care conditions. The intervention with a serious card game (Go Wish) is a patient-centred approach developed to help people discuss their wishes of EOL care and to formalize them in ADs. Compared to previous interventions, it has some major advantages: it is accessible (no literacy barriers), it is specific (it is centred on the needs and wishes about care priorities), and it is adaptable depending on how patients feel ready to engage in such discussions. And most important of all, it is compatible with the Terror Management theory (TMT) that provides explanations on reluctance to write ADs and how to work around this problem. The TMT is a theoretical rationale that posits that death thoughts, occurring during EOL care discussions, operates as barriers by creating an existential anxiety and defence mechanisms. From the TMT perspective, it is possible to reduce the perceived health-related anxiety by helping people to become aware of their own death. This can be achieved by facilitating discussions about EOL preferences and on psychosocial, cultural, and spiritual values of life. The Go Wish intervention focuses on these individual's important life dimensions which could reduce anxiety in the process of ACP and ADs completion and alleviate defensive behaviours present in EOL care.

Primary objective: To test the efficacy of the Go Wish intervention for increasing the proportion of ADs completed in outpatients receiving early stage of palliative care services compared to usual care (i.e. standardized information on ADs).

Secondary objectives: To explore the role that TMT defence mechanisms plays in the process of end-of-life discussions in nurses, patients and relatives (mixed method).

DETAILED DESCRIPTION:
Background and rationale: In Switzerland, only 10% of deaths per year occur suddenly and unexpectedly and about two thirds of people die from an illness after receiving medium to long-term medical care for their life limiting conditions. A large proportion of the population has an invested interest in the process of advance care planning (ACP) for end-of-life care and the use of anticipated directives (ADs). The purpose of ADs is to give people the opportunity to indicate their preferences, beliefs, values or fears to healthcare professionals and choose a surrogate, in case of loss of capacity and discernment.

Despite perceived utility of ADs, interventions to increase rates of legally completed ADs have produced few significant increases in their uptake and use. For instance, literature shows that in Swiss about 5-14 % of adults have completed ADs. Recent research shows that, even when people are informed about ADs, a great majority do not formalise their choices by writing their ADs. This raises questions about how best to encourage patients (passively or actively) to engage in the process of ADs and how health professionals could support them.

Current developments in anticipated decision-making shifted from the traditional completion of ADs towards Advance Care Planning (ACP). This concept is seen as a continuous development of communication between patients, close relatives and health professionals with the aim to define a common orientation for care and treatment. ADs are now seen as part of the ACP process which focused on preferences, goals of care, life-sustaining treatments, palliative options, surrogate decision-making and documentation (as ADs).

Some recent systematic reviews highlight the heterogeneity of ACP interventions, setting stakeholders, designs, measures or outcomes. The efficacy of ACP interventions for different populations, and more specifically in the completion of ADs and the occurrence of end-of-life discussions was shown in some studies. However, it is not clear which elements of ACP are effective and how to best favour the implementation of it in practice. There remains nevertheless, a lack of well-conducted RCTs to evaluate ACP intervention irrespective of the setting. And this needs to be improved by developing intervention programs in the topic and to overcome barriers that might limit engagement in ACP, such as professionals', patients' and close relatives' discomfort with end-of-life issues.

Hospital stays are increasingly being shortened and as a consequence, patients are exposed to a multitude of professionals who may not be in a position to adequately discuss the delicate subject of end-of-life care, due to the priority of providing acute care for many patients. Moreover, when focusing on populations near the end of their lives (life expectancy less than six months), for around 40% of patients, it was too late to initiate ADs (and thus ACP) due to cognitive impairment.

Therefore, it may be beneficial to focus on people in 'early stage of palliative care' such as those with chronic degenerative conditions reducing life expectancy, who receive care outside the hospital setting in their natural environment. Therefore, it is preferable to offer a complex ACP intervention at home, considering this setting as a more optimal place to initiate conversations about end-of-life issues.

Recently, a new research avenue uses "card games" to explore end-of-life issues. These tools are considered as a non-threatening way to start a conversation on end-of-life, but their characteristics, objectives and utilization differ (e.g., "Hello" or "Go Wish").

The "Go Wish" tool shows promise for our population of interest. It is a patient-centred approach to help people to discuss their preferences and options of end-of-life care, to formalize them in ADs and to empower self-determination. It promotes collaborative partnership and shared decision-making with health professionals. It is classified as a serious game and is composed of 36 cards where each card presents a statement that refers to personal needs, values, and beliefs about end-of-life care. The statements have been identified from the literature as particularly important because they correspond to descriptors of "a good death" and they relate to four main dimensions: (a) oneself, (b) care (technical, physical, relational, and spiritual), (c) family and close relatives, and (d) context and organization of end-of-life. Experience with the cards showed good feasibility and acceptability to the different participants it was tested on (nurse, patients and close relatives). The advantage of the Go Wish, compared to the previous mentioned ACP's interventions, is its accessibility (no literacy barriers) and that it is more centred on the needs and wishes of the patient instead of being centred on the disease as the others mentioned above. Another major advantage of this intervention is that patient initiates and guides discussions on themes she/he wants to develop, meaning the patient's own readiness is respected and reflected in her/his engagement in these complex processes such as those defined in the Prochaska's Transtheoretical model. This model proposes five steps relevant to change and is a frequently used theory in ACP. It offers a framework that specifies the different strategies needed at each stage to change attitudes, intentions and behaviours that are implicated in the ACP and ADs process.

Nevertheless this model does not explain the complexity involved with psychological mechanisms of defence that are present in end-of-life thinking such as those experienced by patients, their closes relatives and carers and health professionals when considering ACPs and ADs. Therefore, there is a need to understand people's reluctance to formalize ADs and work around this problem. On another hand, a psychosocial model, the Terror Management Theory (TMT) could offer an explanation. It is a theoretical framework based on the assumption that human individuals, in contrast to all other beings, are confronted with the awareness that they will sooner or later inevitably die. This mixture of the inevitability of mortality as a reality of their lives, coupled with their striving for survival, can produce a paralyzing anxiety or terror that needs to be managed.

TMT seems a framework in which to explore the occurrence of psychological mechanisms described below in end-of-life discussion contexts. A few qualitative studies suggest that getting involved in an ACP process can lead people to prematurely think about their death creating unnecessary anxiety. Because "being diagnosed with a serious illness, receiving or providing medical treatment" reminds people (both professionals and lay people) of their own inevitable mortality, the question arises how best to encourage people engaging in health preferment activities, such as ACP. From the TMT perspective, it is possible to reduce the perceived health-related anxiety by helping people to become aware of their own death by facilitating discussions about end-of-life preferences.

The Go Wish intervention focuses on individual's important life dimensions, which could reduce anxiety in the process of ACP and ADs completion and alleviate defensive behaviours present in end-of-life care.

Objectives: Grounded in the TMT, the efficacy of the Go Whish intervention compared to the standardized information on ADs commonly used in outpatients with progressive chronic illnesses will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Nurses: stable contract, with a diploma in nursing, fluent in French, being able to provide informed consent;
* Patients: at least 18 years old, chronic progressive disease impacting life expectancy, being able to speak, read and understand French, followed by nurses of imad a least once a week, capacity of discernment, being able to provide informed consent;
* Relatives: designed by the patient, at least 18 years old, being able to speak, read and understand French, capacity of discernment, being able to provide informed consent

Exclusion Criteria:

* Nurses: temporary work, refusal to provide informed consent
* Patients: existing ADs, terminal care, existing diagnosis of cognitive disorders or sensory motor impairment documented in the patient file related to memory loss or disturbances of speech that would not allow for a constructive exchange, refusal to provide informed consent;
* Relatives: imad's professional, refusal to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of completed anticipated directives | 6 months after inclusion
  Completion of anticipated directives will be coded "yes" when anticipated directives are written and signed, otherwise it will be coded "no"

SECONDARY OUTCOMES:
Level of anxiety | for patients and relatives: baseline; at three months; for nurses: baseline; at 1, 3 and 12 months
  Level of anxiety will be measured using the validated French version of the Positive and Negative Affect Scale (PANAS). It consists of two 10-item scales to measure mood: positive and negative affect (with two sub-scales: afraid and upset). Items are rated on a 5-points Likert scale.
  A high score on the positive affect scale denotes an optimal state of energy, concentration, and pleasurable engagement whereas a low score reflects sadness and lethargy. A high score on the negative affect scale indicates distress and unpleasant engagement whereas a low score denotes calmness and serenity.
Attitudes towards ADs | baseline; at 1, 3 and 12 months
  For nurses: It will be measured using the validated Knowledge Attitudes and Practice Behaviors Questionnaire (KAP), translated-back translated in French. KAP is 53-item scale composed of five dimensions: (a) demographic and practical characteristics (11 items), (b) knowledge about ADs cares (12 items), (c) attitudes face with ADs (18 items) split up into -beliefs (8 items) - subjective norms (6 items) - control perception (4 items), (d) practices during discussions (4 items), (e) other information on practice (8 items). The questions related to knowledge about ADs cares (12 items) were excluded (not relevant for the research questions). Items are rated on a 5-points Likert scale.
Quality of end of life communication | baseline; at three months
  For patients: Quality of end of life communication between patient and nurse will be measured using the validated "Quality of patient-clinician communication about end-of-life care" (QOC). It is a 19-item scale composed of two subscales: a) global communication competencies of the clinician (7 items) and b) specific competencies determining the quality of the communication about end-of-life care (12 items). Items are rated on a 10-points Likert scale. Translation and back translation procedure will be run.
Patient Empowerment | baseline; at three months
  For patients: Patient empowerment will be measured using the validated French version of the "Health care empowerment questionnaire (HCEQ)". A 10-item scale that evaluates the degree of "empowerment" perceived by the patient with the care received and health services on a 4-point Likert scale.
Quality of life patients | baseline; at three months
  For patients: Quality of life will be measured using the French validated version of the "McGill quality of life revised (MQOL-R)". It is a 14-item scale composed of a four sub scales (plus a general quality of life question (1 item)): physical (3 items), existential (4 items), psychological (4 items) and social (3 items). Items are measured on an 11-points Likert scale.
Quality of life of relatives | baseline; at three months
  For the relatives: quality of life will be measured using the validated French version of World Health Organization Quality of Life (WHOQOL) brief. It is a 26-item scale based on satisfaction questions across four domains of quality of life: physical health (7 items), psychological health (6 items), social relationships (3 items), environment (8 items), and two general questions. Items are rated on a 5-points Likert scale in reference to the last 2 weeks. A percentage rating within each domain was computed with scores ranging from 0 (lowest quality of life) to 100 (highest quality of life) as defined by the instrument use.

CONTACTS AND LOCATIONS:
Overall Officials: Katia Iglesias, PhD, Principal Investigator — HES-SO University of Applied Sciences and Arts of Western Switzerland
Locations (1):
- IMAD, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iglesias K, Busnel C, Dufour F, Pautex S, Sechaud L. Nurse-led patient-centred intervention to increase written advance directives for outpatients in early-stage palliative care: study protocol for a randomised controlled trial with an embedded explanatory qualitative study. BMJ Open. 2020 Sep 20;10(9):e037144. doi: 10.1136/bmjopen-2020-037144. PMID 32958487